CLINICAL TRIAL: NCT00802451
Title: A Study to Evaluate the Relative Bioavailability of Two Mesalamine 4 gm/60 ml Rectal Enema Formulations
Brief Title: Bioavailability Study of Two Mesalamine 4 gm/60 ml Rectal Enema Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10216928
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Bioavailability; Mesalamine
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Drug (Active Comparator)
  Interventions: Drug: Mesalamine
- Reference Drug (Active Comparator)
  Interventions: Drug: Mesalamine

INTERVENTIONS:
Drug: Mesalamine

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of the test formulation of mesalamine suspension rectal enema with the reference formulation in healthy, adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women, 18 to 55 years of age
* weight within +/- 25% for height and weight for body frame
* willing to participate and sign a copy of the informed consent form

Exclusion Criteria:

* recent history of drug or alcohol addiction or abuse
* pregnant or lactating women
* history of allergic response to mesalamine
* evidence of a clinically significant disorder or whose laboratory results were deemed to be clinically significant
* receipt of any drugs as part of a research study within 28 days prior to study dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2003-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence was assessed on the pharmacokinetic variables, Cmax, AUCO-t and AUCO-infinity